CLINICAL TRIAL: NCT06688032
Title: Efficiency Comparison of Jarlsberg- and Norvegia Cheese on Bone Markers, Resting Metabolic Rate, Bone Mineral Density, Muscle Strength and Peak VO2 in Cross-Country Skiers of Both Sexes
Brief Title: Efficacy Comparison of Jarlsberg- and Norvegia Cheese on Bone Markers and Bone Mineral Density in Nordic Skiers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meddoc (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor Emeritus, Meddoc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XCS-Jarlsberg/IIA
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Bone Health; Performance Enhancing Product Use
Keywords: XCS; Bone markers; Cheese; Muscle strength

STUDY DESIGN:
Intervention Model Description: Design and randomization The study was performed as an open randomized stratified parallel group designed trial with two strata. Sex is used as a stratification factor. The two equal sized strata are chosen because of different OED of cheese for women and men, and because the dose-response study previously performed has shown different response in men and women. The participants were equally allocated (1:1) to either Jarlsberg or Norvegia cheese by block randomization.
Masking Description: Blinding was not possible due to the look and tast of the two cheeses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jarlsberg cheese (Active Comparator): Daily oral intake of 75g and 90g Jarlsberg cheese to females and males, respectively
  Interventions: Other: Jarlsberg cheese
- Norvegia cheese (Active Comparator): Daily oral intake of 75g and 90g Norvegia cheese to females and males, respectively
  Interventions: Other: Norvegia

INTERVENTIONS:
Other: Jarlsberg cheese — Jarlsberg cheese contains Propionebacterium freudenreichii (PF) producing the K2-vitamer MK-9(4H) and DHNA in addition to the K2-vitamers found in Norvegia cheese
  Other Names: Oral daily intake of Jarlsberg cheese
  Arms: Jarlsberg cheese
Other: Norvegia — Cheese with different content of K2 vitamers
  Other Names: Oral daily intake of Norvegia cheese
  Arms: Norvegia cheese

SUMMARY:
The study objective consists of the following two aims:

1. Compare the effect of daily intake of Jarlsberg and Norvegia cheese on bonehealth in active Cross Country- and Biathlon skiers of both sexes.
2. Compare the effect daily intake of Jarlsberg and Norvegia cheese in change of the metabolism , Muscle Strength, Muscle Mass and endurace in active Cross Country- and Biathlon skiers of both sexes.

Population and sampling; The study population consists of active skiers of both genders past 17 years of age for females and 18 years for males. The study sample concists of 30 female and 30 male skiers equally randomized to either Jarlsberg or Norvegia cheese for 24 weeks.

Study performance: Blood samples were collected at baseline and every eight week. Metabolism , Muscle Strength, Muscle Mass and endurance were recorded at start and at the end of the study. Diet and exercise volume were recorded and monitored every eight weeks together with daily cheese intake.

DETAILED DESCRIPTION:
1 Objectives

The study objective consists of the following two aims:

i. Compare the effect of daily intake of Jarlsberg and Norvegia cheese in change of the OC level and Carboxylated Osteocalcin(cOC), Bone Mineral Density (BMD), Trabecular bone score (TBS) and other bone markers in active Cross Country Skiers and Biathlon skiers both sexes.

ii. Compare the effect daily intake of Jarlsberg and Norvegia cheese in change of the Resting metabolic rate (RMR), Muscle Strength (MS), LM and Peak VO2 in active Cross-country Skiers and Biathlon Skiers of both sexes.

2: Population and sampling The study population consists of active Cross-country and Biathlon Skiers both sexes past 17 years of age for females and 18 years for males.

4: Study procedure i)Screening: The recruited skiers who fulfilled the inclusion and avoided the exclusion criteria were screened during 1 week. The participating candidates fulfilling the criteria and signed the informed consent form for participation were included. Physical activity and diet registration were performed. The week before the first investigation, the participants were asked to fill in their diet for four days in a data application created for this study. The diet registration was performed and monitored.

ii) First comparison part: The duration of the first comparative part is eight weeks. The XCS will randomly be allocated (1:1) to either daily intake of Jarlsberg cheese or Norvegia cheese for 8 weeks. The daily intake of Jarlsberg® cheese will be the sex-related estimated optimal efficacy dose (OED) for XCS and the comparative dose of Norvegia. The two cheese doses are nearly equal regarding total energy, protein, carbohydrate, fat, and calcium. The trial cheese can be consumed with other food at breakfast, lunch, or other meals during the day. The daily doses of both cheeses will be 5 slices of cheese (75g/day) for females and 6 slices (90g/day) for males The first clinical investigation in the study was take place and is denoted as Day 0. The participants was receive a study identification number and informed not to use other cheese than the one received in the study. During this initial clinical examination, all demographic data, social factors, history of disease and vital signs was recorded. Blood samples was drawn fastening for measurements of Osteocalcin and vitamin K2; Haematological and biochemical variables like HbA1C and Lipids, magnesium, calcium, phosphate, and urea; Collagen (CTX-1) and procollagen (PINP), parathyroid hormone (PTH), and bone specific alkaline phosphatase (BALP); Estradiol and testosterone; LH, FSH and SHBG. Additionally, a DXA with VAT and Bodyfat (BF) investigation was performed. In addition to BMD and TBS, the body composition variables Lean body mass (LM) and Fat free mass (FFM), was measured together with RMR, muscle strength and Peak VO2 before starting the clinical part.

After four weeks the participants meet for the second visit. Blood samples for measurements Osteocalcin and the specific bone turnover markers (BTM) was drawn. The participants were given a new sample of cheese and calcium tablets for the next four weeks and new date for the next visit.

Diet registration for four days was performed in the data application every 8 weeks in the study. The diet registration was monitored by a professional nutritionist.

The last investigation in this first comparative part was take place at week 8. The participants will undergo a common clinical examination like the one performed initially. Blood samples for measurements of Osteocalcin, vitamin K2, and BMT will be taken. Haematological and biochemical variables except for vitamin D, parathyroid hormone (PTH), Estradiol and testosterone; LH, FSH and SHBG will be measured.

iii) Second comparative part: The duration of the second comparative part was 16 weeks and started at study-week 8. The participants received new cheese, and calcium tablets every 4 weeks and met for new clinical examination every 8 weeks.

The first clinical examination the this second comparative part was performed at study-week 16. A diet registration was performed the last week before the visit. A common clinical examination was performed and blood samples for measurements of Osteocalcin, vitamin K2, the specific BTMs, sex hormones and biochemical variables were drawn. The participants were provided new sample of cheese and calcium tablets for four weeks and a date for the next visit.

This visit performed at week 24 was the last clinical examination in the study and equal to the initial study visit. Blood samples were drawn for measurements of Osteocalcin, BTMs, vitamin K2 and biochemical and haematological variables. Sex hormones, muscle strength, Peak VO2, DXA investigation for BMD, TBS and LM, and RMR were measured in the same way as at day 0.

The female participants were interviewed about their menstruation status including menarche length, cycles day and use of hormonal contraception.

iv) Dietary Monitoring: The participants registered their dietary intake in an application at baseline and every 8th week of the study. During the last visit an Eating Disorder Examination Questionnaire- Short, (Prenjak K, et al BMC Psychiatry 2020;20:1-7) derived from EDE-Q © Fairburn and Beglin, 2008 was a part of the interview.

The questions were woven into the anamnestic interview and not as a questionnaire to ensure that the participants do not suffer from disordered eating.

5 Main variables The main variables in this study were the Osteocalcin development, BTMs, RMR and BMD. Supporting variables were muscle strength, LM and Peak VO2 and gender hormones. The vitamin K2 variants MK-7, 8, 9, 9(4H), HbA1C, vitamin D, Ca++, Mg++ and urea, were secondary variables. As safety variables, haematological- and biochemical variables and adverse events (AE) were recorded at each visit. The participants' activity was be continuously recorded.

5: Sample size With a significance level of 5%, a power of 90% and a clinically relevant difference in total osteocalcin increase of one-time SD between the two groups, at least 24 XCSs in each group must be included. By correcting for dropouts during the first part of the study, 30 XCS were included in each group. Totally 60 skiers were recruited for participation.

ELIGIBILITY:
Inclusion Criteria:

* Active Cross-country and Biathlon skiers from 17 years of age for females and 18 years for males.

Exclusion Criteria:

* Eating disorder
* Pregnancy
* Serious gastrointestinal disorder.
* Abnormal liver or kidney function.
* Diabetes
* Suffering from verified cancer.
* Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* Known milk product allergy.
* Suffering from diseases or injuries that disable them to perform VO2 or muscular strength tests.
* Not able to understand information.
* Do not want or not able to give written consent to participate in the study.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
BMD | From baseline to 24 weeks
  Bone Mineral Density

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian School of Sport sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundberg HE, Larsen S, Mathisen TF, Sundgot-Borgen J. Comparison of cheese with and without Propionibacterium freudenreichii subsp. shermanii LMGT 2951 on off-season muscle strength and VO2 max development in Nordic skiers: a randomized clinical trial. J Int Soc Sports Nutr. 2025 Dec;22(1):2566373. doi: 10.1080/15502783.2025.2566373. Epub 2025 Sep 30. PMID 41025612

DOCUMENTS (1):
  • Study Protocol (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT06688032/Prot_000.pdf